CLINICAL TRIAL: NCT01683045
Title: Ablation for the Treatment of Concomitant Atrial Fibrillation in Non-Paroxysmal Patients (ATTAC-AF)
Brief Title: Efficacy and Safety Study of the Estech COBRA® Surgical System to Treat Patients With a History of Irregular Heart Beats
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Endoscopic Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 400-02; ATTAC-AF
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: non-paroxysmal atrial fibrillation; persistent atrial fibrillation; atrial fibrillation; heart palpitations; irregular heart beat; temperature-controlled radiofrequency ablation; radiofrequency energy; TCRF energy; RF energy; epicardial and endocardial lesions; concomitant heart surgery; surgical ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Estech COBRA® Surgical System (Experimental)
  Interventions: Device: The Estech COBRA® Surgical System

INTERVENTIONS:
Device: The Estech COBRA® Surgical System — The Estech COBRA® Surgical System has been designed to create epicardial and endocardial lesions on the heart using temperature controlled radiofrequency (TCRF) ablation with the Estech COBRA surgical probes. Temperature control provides a meaningful endpoint, maintaining tissue at safe yet effective temperatures to produce the desired lesion set. Internal probe cooling and advanced suction helps to ensure reproducible transmural (full-thickness) endocardial or epicardial lesions.
  Other Names: Estech COBRA Cooled™ Surgical Probe; Estech COBRA Adhere™ XL Surgical System; Estech COBRA Adhere™ XL 2 Surgical System; Estech COBRA® Revolution Bipolar Clamp

SUMMARY:
The purpose of this study is to demonstrate that the Estech COBRA Surgical System is an effective treatment for patients with irregular heart beats who are undergoing heart surgery.

DETAILED DESCRIPTION:
The objective of the trial is to demonstrate that the creation of epicardial and endocardial lesions with temperature-controlled radiofrequency (TCRF) ablation applied using the Estech COBRA® Surgical System during concomitant heart surgery is a safe and effective treatment for non-paroxysmal atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in this trial:

1. Subject is scheduled to undergo elective on-pump cardiac surgical procedure(s) for one or more of the following:

   1. Mitral valve repair or replacement,
   2. Aortic valve repair or replacement,
   3. Tricuspid valve repair or replacement, or
   4. Coronary Artery Bypass procedures;
2. Subject has history of a non-paroxysmal form of AF for greater than 3 months and has failed at least one attempt at electrical cardioversion or had a successful attempt at electrical cardioversion but had a recurrence of AF within 30 days of the cardioversion;
3. Age 18 to 80 years old;
4. Left ventricular ejection fraction (LVEF) ≥ 30%;
5. Subject has no contraindications to intraoperative transesophageal echocardiography;
6. Subject has a life expectancy greater than 12 months; and
7. Willing and capable of providing Informed Consent to undergo surgery and participate in all examinations and follow-ups associated with this clinical trial.

A subject is considered to have failed electrical cardioversion if they did not achieve sinus rhythm for at least 30 seconds following the attempted cardioversion.

Exclusion Criteria:

Subjects will be excluded from participating in this trial if they meet any of the following exclusion criteria:

1. History of non-paroxysmal AF less than 3 months or for more than 5 years;
2. History of prior cardiac ablative surgical or catheter-based therapy;
3. Previous cardiac surgery (redo) or other intrapericardial procedures;
4. Class IV NYHA heart failure;
5. Known carotid artery stenosis greater than 80% or previous carotid endarterectomy;
6. Wolff-Parkinson-White syndrome;
7. Need for emergent cardiac surgery (e.g., cardiogenic shock);
8. Untreated hyperthyroidism;
9. Untreated hypothyroidism;
10. Acute pulmonary disease;
11. Electrolyte imbalance;
12. History of myocarditis;
13. Presence of a previously implanted device in or adjacent to the treatment target area that may alter the delivery of therapy (e.g., valvular prosthesis or ring, pacemaker with leads in coronary sinus or internal defibrillator leads);
14. History of pericarditis;
15. Previous left phrenic nerve paralysis;
16. Bullous lung disease;
17. Presence of active endocarditis, or local or systemic infection;
18. Recent myocardial infarction (< 3 months);
19. Renal failure requiring dialysis or hepatic failure or creatinine of >2 mg/dL preoperatively;
20. Antiarrhythmic drug therapy required for the treatment of a ventricular arrhythmia;
21. Preoperative need for an intra-aortic balloon pump or intravenous inotropes;
22. Severe peripheral arterial occlusive disease defined as claudication with minimal exertion;
23. Therapy resulting in compromised tissue integrity including: thoracic radiation, chemotherapy, long term treatment with oral or injected steroids, or known connective tissue disorders;
24. Documented left atrial size of 6 cm or more;
25. History of cerebrovascular disease or accident, including stroke or transient ischemic attack (TIA) within 6 months prior to enrollment;
26. Known contraindication to anticoagulant therapy or inability to comply with anticoagulant therapy;
27. Pregnancy, planned pregnancy (females of childbearing potential must have a negative pregnancy test prior to enrollment and agree not to become pregnant during the trial) or breastfeeding;
28. Forced expiratory volume in 1 second less than 30% of predicted value or need for home oxygen therapy; or
29. Surgical management of hypertrophic obstructive cardiomyopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | The primary efficacy endpoint will be assessed following the blanking interval through Month 12.
  Proportion of subjects that achieve procedural and therapeutic success. Procedural success is defined as the performance of the protocol specified lesions with the designated devices. Therapeutic success is defined as freedom from AF, AFL (atrial flutter) and AT (atrial tachycardia, not including sinus tachycardia) following the blanking interval through Month 12.
Primary Safety Endpoint | The primary safety endpoint will be assessed within 30 days of the procedure or hospital discharge, whichever is later.
  A composite safety endpoint consisting of the proportion of subjects that experience one or more of the following early onset (i.e., within 30 days of the TCRF ablation procedure or hospital discharge, whichever is later) serious adverse events (SAEs):
  * Cardiac death;
  * Stroke and transient ischemic attack (TIA);
  * Myocardial infarction (MI);
  * Excessive bleeding; or
  * Atrioesophageal fistula.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | The secondary efficacy endpoints will be assessed following the procedure through the 12 month follow-up visit.
  The secondary efficacy endpoints include:
  * Proportion of subjects that achieve bilateral pulmonary vein conduction block.
  * AF burden at 6 and 12 months based on the proportion of time a subject is in AF (% of 24 hours) from the 24-hour continuous ECG monitor.
Secondary Safety Endpoint | The secondary safety endpoints will be assessed up to 3 years post procedure.
  The proportion of subjects with acute onset post-surgical symptomatic diaphragmatic paralysis that is still present at the Month 12 follow-up visit.
  The proportion of subjects reporting one or more SAEs for each follow-up interval. The intervals will include the period from:
  * the surgical procedure for the surgical TCRF ablation through the Day 30 follow-up visit;
  * the Day 30 follow-up visit through the Month 3 follow-up visit;
  * the Month 3 follow-up visit through the Month 6 follow-up visit; and
  * the Month 6 follow-up visit through the Month 12 follow-up visit. Additionally, the proportion of subjects reporting one or more SAEs annually for years 2 and 3 post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David K Swanson, Ph.D., Principal Investigator — Endoscopic Technologies, Inc
Locations (13):
- United States (13):
  - Banner Good Samaritan Medical Center, Mesa, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - North Shore Univ. Health System, Evanston, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - The Univ. of Kansas Hospital, Kansas City, Kansas
  - Univ. of Michigan Cardiovascular Center, Ann Arbor, Michigan
  - Mayo Clinic / St. Mary's Hospital, Rochester, Minnesota
  - Lenox Hill Hospital / North Shore-LIJ Health System, New York, New York
  - Mohawk Valley Heart Institute / St. Elizabeth Medical Center, Utica, New York
  - Sisters of Charity, Providence Hospital, Columbia, South Carolina
  - Fairfax Hospital, Department of Cardiovascular and Thoracic Surgery, Falls Church, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin